CLINICAL TRIAL: NCT06566664
Title: Peripheral Neurostimulation for Nerve Block Placement
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jean-Louis Horn, Professor of Anesthesiology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 76523
Record Dates: First submitted 2024-08-07; First posted 2024-08-22 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-11

CONDITIONS: Pain Syndrome; Pain Management
Keywords: peripheral nerve block; neurostimulation
MeSH Terms: conditions — Somatoform Disorders; Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Ultrasound-guided brachial plexus block with peripheral nerve stimulation (Experimental): Patients will receive a brachial plexus catheter with ultrasound guidance as per standard of care, with additional use of the B. Braun HNS 12 nerve stimulator during the loading dose of local anesthesia to maintain a gentle twitch.
  Interventions: Device: B Braun HNS 12 nerve stimulator
- Ultrasound-guided brachial plexus block without peripheral nerve stimulation (Sham Comparator): Patients will receive the brachial plexus catheter in the same way the first arm would, and the B Braun nerve stimulator will be placed in the same way, but the ground electrode will not be connected to the patient.
  Interventions: Device: B Braun HNS 12 nerve stimulator sham control

INTERVENTIONS:
Device: B Braun HNS 12 nerve stimulator — Nerve stimulator that is traditionally used for nerve localization during block placements.
  Arms: Ultrasound-guided brachial plexus block with peripheral nerve stimulation
Device: B Braun HNS 12 nerve stimulator sham control — Stimulator will be placed and turned on, but the grounding electrode will not be connected to prevent nerve stimulation.
  Arms: Ultrasound-guided brachial plexus block without peripheral nerve stimulation

SUMMARY:
Peripheral nerve blocks are routinely used and highly successful for intra-operative anesthesia and post-operative pain management. Nerve blocks are guided using either neurostimulation as a means to localize the right nerve or by ultrasound guidance or combining the 2 methods. The purpose of this study is to assess whether electrical stimulation improves nerve block quality, beyond its simple purpose of nerve localization.

DETAILED DESCRIPTION:
The investigators wish to understand how electrical stimulation can affect local anesthetic disposition when performing a peripheral nerve block.

By studying this subject, the investigators open possibilities for improvement on many levels:

increasing the efficacy of the nerve block allows for a reduced onset time, reduced incidence of incomplete block and prolonged duration of the local anesthetics. This allows for patients to fully benefit from the analgesic properties of the nerve block, allows for a decrease in delays for the operating room readiness, and a decrease in the amount of medication needed for a successful nerve block. This will decrease side effects and risks of the nerve blocks. Overall better post-surgical pain control may decrease risks for developing chronic post-operative pain, a major post-operative complication.

The results of this study will open the door to novel approaches to manage acute post-operative pain.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective upper limb surgery with a planned brachial plexus nerve block

Exclusion Criteria:

* Under 18 years old
* ASA score above III
* Chronic pain condition with daily milligrams of morphine equivalent > 30
* Poorly controlled psychiatric condition
* Coagulopathy
* Active infection
* Moderate, severe or progressing neuropathy
* COPD/Chronic oxygen user
* Pregnancy
* Incarceration
* Unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Onset of sensory block | Within 1 hour after the block placement
  Determining time when patient experience first symptoms of local anesthetic action on the upper trunk distribution (median or musculo cutaneous nerve)

SECONDARY OUTCOMES:
Onset of motor block | Within 1 hour after the block placement
  Determining time when patient start loosing strength at the musculo cutaneous nerve (biceps brichialis muscle)
Duration of sensory block | up to 7 days after surgery
  Time after surgery at which the patient recovers first sign of sensory function
duration of motor block | up to 7 days after surgery
  Time after surgery at which the patient recovers a biceps brachialis function
When patient experience first pain | up to day 7 post operatively
  Time after surgery at which the patient experience first sign of pain at the surgical site
Time of first opioid taken | within the first 7 days after surgery
  When the first opioid was taken
Opioid usage at day 1 | at post operative day 1
  Milligram of morphine equivalent
opioid usage assessment at day 7 | Within the Post operative day 1 and 7
  Milligram of morphine equivalent taken
Opioid usage assessment at day 28 | usage between post operative day 7 and 28
  milligram of morphine equivalent assess at day 28
Last opioid usage after day 28 | Assessment within 1 year
  When was the last day of opioid usage
Amount of opioid usage after 28 days | 28 days to 1 year after surgery
  Milligram of morphine equivalent use weekly after 28 days
Patient satisfaction | At Post Operative day 7, 28 and 1 year
  Assessing patient's satisfaction, using the standardized -Quality of Recovery 15- at post operative day 7, 28 and 1 year. Each item count on a 0-10 scale where O is worse and 10 is best PART A How have you been feeling in the last 24 hours? (0 to 10, where 0 = none of the time [poor] and 10 = all of the time [excellent] Q.1 Able to breathe easily Q.2 Been able to enjoy food Q.3 Feeling rested Q.4 Have had a good sleep Q.5 Able to look after personal toilet and hygiene unaided Q.6 Able to communicate with family or friends Q.7 Getting support from hospital doctors and nurses Q.8 Able to return to work or usual home activities Q.9 Feeling comfortable and in control Q.10 Having a feeling of general well-being PART B Have you had any of the following in the last 24 hours? (10 to 0, where 10 = none of the time [excellent] and 0 = all of the time [poor]) Q.11 Moderate pain Q.12 Severe pain Q.13 Nausea or vomiting Q.14 Feeling worried or anxious Q.15 Feeling sad or depressed
General satisfaction | at post operative day 7, 28 and 1 year
  General satisfaction on a scale from 1-5 (extremely unsatisfied, unsatisfied, neutral, satisfy, extremely satisfied)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University Hospital, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No